CLINICAL TRIAL: NCT01141166
Title: A Randomised Controlled Trial on Falls and Malnutrition Prevention in the Community in 85 Year Old Subjects
Brief Title: Octabaix Intervention Study
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Collaborators: Preventive Services and Health Promotion Research Network (Other)
Responsible Party: Cecíla Borau, Jordi Gol i Gurina Foundation
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AFF2191
Record Dates: First submitted 2010-04-14; First posted 2010-06-10 (Estimated); Last update posted 2010-06-10 (Estimated); Status verified 2010-06

CONDITIONS: Falls; Malnutrition
Keywords: ELDERLY; NUTRITION
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Who Masked: Participant, Care Provider

ARMS (1):
- nutritional and physical rehabilitation plan (Experimental)
  Interventions: Behavioral: nutritional and a rehabilitation plan.

INTERVENTIONS:
Behavioral: nutritional and a rehabilitation plan. — The intervention consisted of recommendations to the subject and their primary physician, and others providers, telephone calls of a nutritional and a rehabilitation plan.

SUMMARY:
Objective: To determine the effectiveness of an individual multifactorial intervention on falls and undernutrition risk in very older people in the community.

DETAILED DESCRIPTION:
Design: Randomized, controlled trial.

Method: Three hundred and twenty eight people born in 1924, after recruitment will be followed for a three year period. Subjects received two in-home visits from a trained nurse or physicians who assessed falls and nutritional risk factors using an algorithm.

The intervention consisted of recommendations to the subject and their primary physician, and other providers, telephone calls, and exercise and nutritional plan. Control subjects received a general primary care assessment.

Measurements: the primary outcome were rate of falls and rate of undernourished risk. Secondary outcomes included different geriatrics characteristics.The outcomes of this study will provide important new information to reduce the incidence of falls and the risk of undernutrition of this population by intervention. Significant differences are not expected according to social-demographics sex and other factors, but they are expected by other obtained factors and indices that could allow to detection of octogenarian people with great risk of deterioration in just a short time.

ELIGIBILITY:
Inclusion Criteria:

* Subjects born in 1924 of one of the 7 participating health centers and noninstitutionalized

Exclusion Criteria:

* Institutionalized

Ages: 85 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 328 (Estimated)
Dates: Start 2009-01; Primary Completion 2011-04 (Estimated)

PRIMARY OUTCOMES:
Rate of falls and rate of undernutrition risk as MNA < 23,5
  Nutritional risk was evaluated by the MNA questionnaire

SECONDARY OUTCOMES:
Different geriatrics characteristics
  Functional, cognitive and nutritional status and social risk were assessed by instruments currently used in geriatric practice. Functional status was measured using the BI (Mahoney and Barthel, 1965) for the basic ADL, and the Lawton index (LI) (Lawton and Brody, 1969). Cognitive function was measured by the Spanish version (MEC) (Lobo et al., 1999) of the MMSE. Comorbidity by the Charlson comorbidity index (CCI)and the others.

CONTACTS AND LOCATIONS:
Locations (1):
- Assumpta Ferrer Feliu, Sant Feliu de Llobregat, Barcelona, Spain

REFERENCES:
- [Derived] Badia T, Formiga F, Ferrer A, Sanz H, Hurtos L, Pujol R. Multifactorial assessment and targeted intervention in nutritional status among the older adults: a randomized controlled trial: the Octabaix study. BMC Geriatr. 2015 Apr 11;15:45. doi: 10.1186/s12877-015-0033-0. PMID 25887312
- [Derived] Ferrer A, Formiga F, Sanz H, de Vries OJ, Badia T, Pujol R; OCTABAIX Study Group. Multifactorial assessment and targeted intervention to reduce falls among the oldest-old: a randomized controlled trial. Clin Interv Aging. 2014 Feb 25;9:383-93. doi: 10.2147/CIA.S57580. eCollection 2014. PMID 24596458